CLINICAL TRIAL: NCT06104111
Title: Investigating the Mechanisms of Epigenetic Memory at the Example of the Responsiveness of Human Immune Cells to Vitamin D
Brief Title: Epigenetic Memory of Vitamin D Supplementation
Acronym: VitDPAS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Polish Academy of Sciences (Other)
Responsible Party: Principal Investigator, Carsten Carlberg, ERA chair of nutrigenomics, Polish Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0001
Record Dates: First submitted 2023-10-19; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Immune System Diseases; Infections; Healthy Lifestyle
Keywords: Vitamin D; Epigenome; Transcriptome
MeSH Terms: conditions — Immune System Diseases; Infections | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D3 (cholecalciferol) (Experimental): 1000 IU vitamin D3 (cholecalciferol)/kg body mass will be taken in form of individual number of pills (4000 IU each, e.g. 20 pills for a person of 80 kg) in the morning together with a breakfast at days 0, 28 and 56
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 bolus at days 0, 28 and 56. Blood samples taken at days 0, 1, 28, 29, 56, 57 ad 84
  Other Names: Cholecalciferol

SUMMARY:
The investigators will study the mechanistic details of dietary programming of the epigenome at the example of epigenetic programming of primary human immune cells with the micronutrient vitamin D3. They will follow a small number of healthy adult volunteers individually over time while measuring per individual a large number of molecular and dynamic parameters that will be used for mechanistic modeling. The main hypothesis of the investigators is that nutritional components, such as vitamin D3, have a direct effect on the epigenome of the different cell types of the immune system. Using complementary in vivo, in vitro and in silico approaches, they will investigate the mechanistic basis of this dietary epigenetic programming process and how it creates memory.

DETAILED DESCRIPTION:
Exposure to dietary molecules during adulthood creates an epigenetic memory in immune cells affecting disease risk in later years of life. Many nutritional molecules have a direct effect on the human genome and/or epigenome, since they (or their metabolites) activate transcription factors or chromatin modifiers. This process is the mechanistic basis of the discipline nutrigenomics. Thus, the daily diet of humans leads to changes in the transcriptome and epigenome of many tissues and cell types. In this way, many physiological functions of the human body, such as a well-responding immune system, are influenced by diet. Some of these effects are not only transient but may lead to persistent changes of the epigenome in many different tissues. However, the mechanistic details of this dietary programming of the epigenome are not well understood. Therefore, in this study, the investigators will study this process at the example of epigenetic programming of primary human immune cells with the micronutrient vitamin D3. They will use the approach to follow a small but sufficient number of healthy adult volunteers (based on power calculation of self-controlled longitudinal studies) individually over time while measuring per individual a large number of molecular and dynamic parameters that will be used for mechanistic modeling, instead of investigating only few parameters from a large number of participants for statistical modeling. The main hypothesis of the investigators is that nutritional components, such as vitamin D3, have a direct effect on the epigenome of the different cell types of the immune system. Using complementary in vivo, in vitro and in silico approaches, they will investigate the mechanistic basis of this dietary epigenetic programming process and how it creates memory.

ELIGIBILITY:
Inclusion Criteria:

-Healthy adult (18-65 years)

Exclusion Criteria:

* Smoker
* BMI > 28 kg/m2
* History of kidney stones, renal failure or dialysis, hypercalcemia, hypo- or hyperparathyroidism, severe liver disease (cirrhosis), or sarcoidosis or other granulomatous diseases, such as active chronic tuberculosis or Wegener's granulomatosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-14 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Vitamin D-induced changes in the epigenome of PBMCs describing the individual -specific vitamin D response index of the study participants | 3 months
  A bolus of vitamin D3 (monthly dose, taken once a month in three repeats) will change the epigenome (and transcriptome) of PBMCs of the study participants in an individual-specific way. These measurements will allow to distinguish the molecular response of the study participants, in order to segregate them into high, mid and low responders to vitamin D. This classification will lead to individual-specific recommendations for daily vitamin D3 supplementation in following winters. Moreover, the molecular investigations will allow a better understanding of the molecular mechanisms of vitamin D responsiveness

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Animal Reproduction and Food Research, Olsztyn, Poland

IPD SHARING:
Plan to Share IPD: No